CLINICAL TRIAL: NCT01922973
Title: Effect of Fasting on Ghrelin and Growth Hormone in Healthy Young and Older Adults
Status: Completed | Type: Observational
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Michael Thorner, MD, Professor of Medicine, University of Virginia
Other Study IDs: 10619
Record Dates: First submitted 2013-08-12; First posted 2013-08-14 (Estimated); Last update posted 2013-08-14 (Estimated); Status verified 2013-08

CONDITIONS: Aging
Keywords: ghrelin; growth hormone; aging; normal volunteers
MeSH Terms: interventions — Angptl4 protein, mouse

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- normal men and women: normal volunteers: young and older men and women studied under fed and fasting (62.5h) conditions with frequent blood sampling for ghrelin and related hormones
  Interventions: Other: Fasting

INTERVENTIONS:
Other: Fasting — normal volunteers fast from food on one occasion for 62.5 h; on another occasion fed 3 meals

SUMMARY:
The overall objective of this study is to determine the extent to which circulating ghrelin levels (total and bioactive ghrelin) are regulated by nutritional state and age.

DETAILED DESCRIPTION:
Normal volunteers: young and older men and women studied under fed and fasting (total 62.5h) conditions, frequent blood sampling for ghrelin and other related hormones

ELIGIBILITY:
Inclusion Criteria:

Healthy young (ages 18-30) and older (ages > 60) men and women with a body mass index (BMI) of <35 kg/m2. Young and older subjects will be matched for BMI.

Exclusion Criteria:

1. A history of coronary artery disease, congestive heart failure, peripheral vascular disease, diabetes mellitus, significant hypertension (BP >180 systolic or >100 diastolic at rest); renal, hepatic, pulmonary disease; untreated hypothyroidism, untreated hyperthyroidism; history of seizure disorder; history of malignancy (other than some skin cancers), history of active chronic infections (e.g., HIV, tuberculosis): abnormal screening laboratory tests. This information will be obtained through the use of screening labs, history and physical exam and the medical record. See the GCRC protocol for details of the labs.
2. Hematocrit < 41% men, < 38% women
3. History of daily tobacco use within past 3 months
4. Chronic alcohol abuse
5. Recent weight change of > 10 pounds in last 3 months
6. Strenuous exercise for average of more than 60 min/day
7. Investigational drug within past 6 weeks
8. Any history of major psychosis, severe depression, anorexia nervosa
9. Transmeridian travel within 2 weeks prior to or during study -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: normal volunteers
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2003-05; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Ghrelin concentration | 24-h mean

CONTACTS AND LOCATIONS:
Overall Officials: Michael O Thorner, MD, Principal Investigator — University of Virginia